CLINICAL TRIAL: NCT04153006
Title: Sample and Method Comparison With Minicare® Point-of-care Device for Cardiac Troponin I Assay at the Emergency Department.
Brief Title: Comparison of Fingerstick Versus Venous Sample for Troponin I.
Status: Completed | Type: Observational
Sponsor: VieCuri Medical Centre (Other)
Collaborators: Siemens Healthcare Diagnostics Inc (Industry); Minicare® B.V. (Unknown)
Responsible Party: Principal Investigator, Braim Rahel, Principal investigator/Cardiologist, VieCuri Medical Centre
Other Study IDs: Study number 478; NL70186.096.19 (Other: ToetsingOnline/CCMO)
Record Dates: First submitted 2019-11-01; First posted 2019-11-06 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Chest Pain; Myocardial Infarction; Myocardial Ischemia; Heart Attack
Keywords: Troponin; Point-of-care; Minicare
MeSH Terms: conditions — Chest Pain; Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain patients: Patients who are admitted to the cardiac ED because of chest pain for ruling out acute coronary syndrome by troponin analysis are eligible for participation.
  Troponin analysis will be performed according to standard protocol (0-1h protocol). From every included patient capillary blood samples and an extra venous blood sample will be drawn to evaluate HS cTnI levels obtained with the POC instrument and central laboratory (CL).
  Interventions: Device: POC troponin analysis.

INTERVENTIONS:
Device: POC troponin analysis. — Point-of-care (POC) high sensitive troponin I (HS cTnI) analysis in whole blood, plasma and capillary whole blood with the Minicare® device.

SUMMARY:
This study is a prospective, observational, cohort study aiming to compare point-of-care high-sensitive troponin I testing from different sample types with central laboratory (CL) HS cTnI plasma samples.

A registry of all included patients and their troponin results (POC, CL and HS cTnT) will be made to compare these testing methods.

DETAILED DESCRIPTION:
Point-of-care (POC) troponin testing, defined as laboratory testing near a patient location with rapid availability of results, has attracted much interest in the emergency department setting (ED) and seems feasible. These devices might enable earlier decisions, reduce stay at the ED and improve patient flow. While an elevated troponin in patients with suspected acute coronary syndrome (ACS) confirms diagnosis and initiates adequate treatment, ruling out ACS aids in proper patient dismissal. A next step could be ruling out myocardial infarction by the general practitioner (GP) or fast responder using an on-site POC troponin test. However, drawing venous blood might not be easily available to every GP, especially not during peak hours. The Minicare cTnI is a bedside system which requires capillary blood, venous whole blood or plasma. The results of the troponin will be given within 10 minutes. It is a very sensitive troponin test, the most clinically sensitive available POC for c-Troponin. Currently Minicare prepares for a high sensitive troponin analysis targeting a reliable result within an hour after onset of chest pain. The objective of this study is to determine if high sensitive troponin testing by Minicare (POC HS cTnI) has the same analytical performance as standard high sensitivity troponin I testing in our central hospital laboratory ( CL HS cTnI ARCHITECT immunoassay analyzer, Abbott).

ELIGIBILITY:
Inclusion criteria:

• Patients 18 years or older with chest pain suspected of ACS.

Exclusion criteria:

* ST elevation myocardial infarction and out of hospital cardiac arrest.
* Patients with sudden onset tachycardia and a frequency of 110 bpm or higher (supraventricular or ventricular)
* Patients who are hemodynamically unstable or in which an acute non-coronary diagnosis is suspected, e.g. pulmonary embolism, thoracic aortic dissection etc.
* Patients recently already admitted for the same set of symptoms at a previous healthcare institution before being transferred to the participating clinical site.
* Patients not willing or not able to provide informed consent due to their medical condition as judged by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presented at our cardiology ED are eligible for inclusion if they are 18 years or older and suspected of having an ACS based on history, examination, and ECG.
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
Method and sample comparison | 30 days
  The primary objective is to compare the analytical performance (method and sample comparison) of Minicare® high sensitive troponin I testing (POC, different sample types) and conventional venipuncture troponin I test in our central hospital laboratory (CL) with the Abbott Architect.
  This comparison will comprise:
  * Minicare® POC (different sample types) vs conventional HS cTnI CL test (Method comparison)
  * Minicare® capillary vs. Minicare® venipuncture and vs. Minicare® plasma (Sample comparison)
  The analyses linked to the primary objectives are:
  * The agreement between POC (three sample types) and CL testing by using the Bland-Altman method.
  * The agreement between different POC sample types by using the Bland-Altman method.
  The primary objective will be achieved by taking capillary and (an extra) venous blood samples (one per timepoint) from every patient presenting at the cardiac ED with chest pain suspected for ACS.

SECONDARY OUTCOMES:
Major adverse cardiac event (MACE) | 30 days
  MACE is is defined as a composite of cardiac death and myocardial infarction.
Final patients diagnoses. | 30 days
  To compare final patients diagnosis (ACS vs. no ACS) and treatment based on POC venous troponin testing versus CL plasma troponin I testing versus HS cTnT plasma testing (regular patient care).
Overview baseline characteristics. | 30 days
  To create an overview of baseline characteristics of the population.
Linear regression and Pearson's correlation. | 30 days
  * The relationship between POC (three sample types) and CL by linear regression and Pearson's correlation.
  * The relationship between POC sample types by linear regression and Pearson's correlation.
Fals-positive and fals-negatives. | 30 days
  To compare the proportion of false positive and false negative results between the different POC samples and if there is a significant difference.
Safety analysis of POC troponin. | 30 days
  To create an overview of the sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV) of POC and standard laboratory troponin I testing.

CONTACTS AND LOCATIONS:
Overall Officials: Braim Rahel, Dr., Principal Investigator — Viecuri MC
Locations (1):
- Viecuri MC, Venlo, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided